CLINICAL TRIAL: NCT00209209
Title: Efficacy of Maintenance Therapy With Rituximab After Induction Chemotherapy (R-CHOP vs. R-FC) for Elderly Patients With Mantle Cell Lymphoma Not Suitable for Autologous Stem Cell Transplantation
Brief Title: Induction Chemotherapy (R-CHOP Vs. R-FC) Followed by Interferon Maintenance Versus Rituximab Maintenance in MCL
Acronym: MCLelderly
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Mantle Cell Lymphoma Network (Other)
Collaborators: German Low Grade Lymphoma Study Group (Other); Lymphoma Study Association (Other); HOVON - Dutch Haemato-Oncology Association (Other); Nordic Lymphoma Group (Network)
Responsible Party: Principal Investigator, Prof. Dr. M. Dreyling (co-chairman), Professor of Medicine, European Mantle Cell Lymphoma Network
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCL2004-1
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Lymphoma, Mantle-Cell
Keywords: Lymphoma, Mantle-Cell; Elderly patients; Chemotherapy; Maintenance therapy; C04.557.386.480.300.725.500; C15.604.515.569.480.300.725.500; C20.683.515.761.480.300.725.500
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; fludarabine; Interferon-alpha; R-CHOP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): 1. randomisation: R-CHOP
  2. randomisation: IFN maintenance
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Interferon-alpha; Drug: pegylated formula Interferon-alpha 2b; Procedure: chemotherapy: R-CHOP; Procedure: Interferon maintenance
- 2 (Experimental): 1. randomisation: R-FC
  2. randomisation: Rituximab maintnenance
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Fludarabine; Procedure: chemotherapy: R-FC; Procedure: Rituximab maintenance

INTERVENTIONS:
Drug: Rituximab — antibody
Drug: Cyclophosphamide — chemotherapy
Drug: Doxorubicin — chemotherapy
  Arms: 1
Drug: Vincristine — chemotherapy
  Arms: 1
Drug: Prednisone — coricosteroide
  Arms: 1
Drug: Fludarabine — chemotherapy
  Arms: 2
Drug: Interferon-alpha — cytokine
  Arms: 1
Drug: pegylated formula Interferon-alpha 2b — cytokine
  Arms: 1
Procedure: chemotherapy: R-CHOP — immuno-chemotherapy
  Arms: 1
Procedure: chemotherapy: R-FC — immuno-chemotherapy
  Arms: 2
Procedure: Interferon maintenance — cytokine
  Arms: 1
Procedure: Rituximab maintenance — antibody
  Arms: 2

SUMMARY:
The aim of this study is to answer the following independent questions in the treatment of mantle cell lymphomas:

* Can rituximab-fludarabine, cyclophosphamide (R-FC) improve the reduction of lymphoma mass compared to rituximab-cyclophosphamide, doxorubicin, vincristine, prednisone (R-CHOP) and so become a new standard for initial cytoreductive therapy?
* Can maintenance with rituximab substitute the interferon maintenance and even improve the progression free survival in patients after successful initial cytoreductive therapy?

DETAILED DESCRIPTION:
This study investigates two independent questions in the treatment of elderly patients with mantle cell lymphomas:

1. To test in elderly patients with advanced mantle cell lymphoma, whether rituximab plus a combination of fludarabine with cyclophosphamide (6 FC cycles) results in a higher reduction of lymphoma mass measured by the percentage of CR than rituximab combined with the standard chemotherapy scheme (8 CHOP cycles).
2. To compare maintenance therapy with rituximab with maintenance with interferon-alpha or pegylated interferon for progression free survival, after 2 different regimens of induction chemo-immunotherapy in elderly patients with mantle cell lymphoma.

This study will be performed as a prospective, randomized, open-label multicenter phase III trial. All patients will be randomized for an initial cytoreductive therapy with R-FC or R-CHOP.

The parameter for the comparison of R-FC and R-CHOP will be the percentage of complete remissions after initial cytoreductive therapy. According to the known results of R-FC and R-CHOP in lymphoma therapy, a relevant difference between R-CHOP and R-FC in the overall response rates is not expected. For both therapies an overall response rate of about 90% is expected. Since it is well known that the prognosis of patients who do not reach at least a PR in the initial therapy is very poor, it will be also necessary to control this parameter during the study. If an unexpected relevant difference in the overall response rates is observed during the study, the initial randomisation should be stopped and all patients should be assigned to the superior therapy. In this case the CR rates will not be important for the choice of the initial therapy. If no relevant differences in the overall response rates are observed, a one sided Fisher test will be performed at the end of the recruitment to test whether the rate of CR's after R-FC is significantly improved compared to R-CHOP.

The statistical parameters for controlling the overall response rates and for testing the CR rates are chosen in the following way: The working significance level for all statistical evaluations in this part of the study will be set to alpha=0.05. The expected CR rate after R-CHOP is according to the observations about 50%; a clinical relevant improvement by R-FC would be a CR rate of 65%. Such an improvement should be detected by the one sided Fisher test with a power of about 95%. According to these parameters about 246 observations for each treatment would be necessary. To control the overall response rates, a difference of 85% to 95% will be clinically so relevant that initial randomisation should be terminated with a probability of about 95%. Overall response rates will be controlled by a restricted sequential procedure.

Patients achieving at least a partial remission after R-FC or R-CHOP will be randomised for interferon maintenance versus rituximab maintenance in order to evaluate the impact of maintenance therapy in progression free survival.

The improvement expected by the new maintenance with rituximab for progression free survival can be expressed by reduction of relative risk (rr). Since a risk reduction to 60% was observed for indolent lymphomas by interferon maintenance, this seems to be a clinical relevant improvement for the new maintenance therapy. For a working significance level alpha=0.05 and a power of 95% the number of events (relapse or death) necessary for a two sided fixed sample trial is about 200. During this study the progression free survival in patients after successful initial therapy will be monitored by an equivalent restricted sequential procedure with a maximum number of 240 observation.

In order to evaluate the impact of initial therapy and maintenance therapy on overall survival in this patients, a total follow up of about 15 years for this study is expected.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven mantle cell lymphoma according to the World Health Organization (WHO) classification, preferably confirmed by central pathology review before entering the study
* Clinical stage II, III or IV
* Previously untreated patients
* Above the age of 65 years and older or patients at the age between 60 and 65, if not eligible for high dose chemotherapy
* WHO performance grade 0, 1 or 2
* Informed consent according to International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use/European Union Good Clinical Practice (ICH/EU GCP) and national/local regulations
* Measurable disease. If, for example only bone marrow (BM) infiltration, patients can only undergo a second randomization if a CR is obtained.

Exclusion Criteria:

* WHO performance of 3 or more
* Known anti-murine antibody (HAMA) reactivity or known hypersensitivity to murine antibodies
* Leukocytes <2.0x 10^9/l or thrombocytes <100x 10^9/l, unless clearly related to mantle cell lymphoma (MCL) bone marrow infiltration
* Patients previously treated for lymphoma
* Patients without measurable lesions; if, for example only bone marrow infiltration, patients may be included, but can only undergo a second randomization in case of a CR
* Patients with stage I disease
* Patients with central nervous system involvement
* Patients with a history of autoimmune hemolytic anaemia or autoimmune thrombocytopenia
* Patients with serious cardiac disease (uncontrolled arrhythmias, unstable angina, severe congestive heart failure)
* Patients with serious pulmonary, neurological, endocrinological or other disorder interfering with full dosing of CHOP or FC chemotherapy
* Liver enzymes >3x normal or bilirubin >2.5x normal (not due to lymphoma)
* Creatinine >2x normal value, corrected for age and weight (not due to lymphoma)
* Patients with unresolved hepatitis B or C infection or known HIV positive infection
* Uncontrolled infection
* Patients with a serious depression that needed therapy within the last 5 years
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Concomitant or previous malignancies other than basal cell or squamous cell skin cancer, in situ cervical cancer and other cancer for which the patient has been disease-free for at least 5 years

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Estimated)
Dates: Start 2004-01-14 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
First randomisation: Reduction of lymphoma mass measured by the complete remission (CR) rate
Second randomisation: progression-free survival after end of initial chemotherapy

SECONDARY OUTCOMES:
Survival after registration / first randomisation / second randomisation
Survival after start / end of initial therapy
Time to treatment failure after start of initial therapy
Progression free survival after registration / first randomisation / second randomisation
Side-effects of initial therapy
Side-effects of maintenance therapy

CONTACTS AND LOCATIONS:
Overall Officials: Hanneke C. Kluin-Nelemans, PhD, Principal Investigator — University Hospital Groningen, Dept. of Hematology; Martin Dreyling, PhD, Study Chair — University Hospital Grosshadern/LMU, Dept. of Medicine III
Locations (7):
- General University Hospital, 1St Department of Medicine, Prague, Czechia
- Nordic Lymphoma Group, Copenhagen, Denmark
- Groupe D´Etudes des Lymphomes De l´Adulte (GELA), Paris, France
- German Low Grade Study Group (Glsg), Munich, Germany
- Ospedale Ferratotto, Divisione Di Ematologia, Catania, Italy
- HOVON - Dutch Haemato-Oncology Association (HOVON-Datacenter), Rotterdam, Netherlands
- The Maria Sklodowska Memorial, Cancer Center - Inst. of Oncology, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kluin-Nelemans HC, Hoster E, Hermine O, Walewski J, Trneny M, Geisler CH, Stilgenbauer S, Thieblemont C, Vehling-Kaiser U, Doorduijn JK, Coiffier B, Forstpointner R, Tilly H, Kanz L, Feugier P, Szymczyk M, Hallek M, Kremers S, Lepeu G, Sanhes L, Zijlstra JM, Bouabdallah R, Lugtenburg PJ, Macro M, Pfreundschuh M, Prochazka V, Di Raimondo F, Ribrag V, Uppenkamp M, Andre M, Klapper W, Hiddemann W, Unterhalt M, Dreyling MH. Treatment of older patients with mantle-cell lymphoma. N Engl J Med. 2012 Aug 9;367(6):520-31. doi: 10.1056/NEJMoa1200920. PMID 22873532
- [Derived] Hoster E, Delfau-Larue MH, Macintyre E, Jiang L, Stilgenbauer S, Vehling-Kaiser U, Salles G, Thieblemont C, Tilly H, Wirths S, Feugier P, Hubel K, Schmidt C, Ribrag V, Kluin-Nelemans JC, Dreyling M, Pott C; European MCL MRD Working Group and the European MCL Network. Predictive Value of Minimal Residual Disease for Efficacy of Rituximab Maintenance in Mantle Cell Lymphoma: Results From the European Mantle Cell Lymphoma Elderly Trial. J Clin Oncol. 2024 Feb 10;42(5):538-549. doi: 10.1200/JCO.23.00899. Epub 2023 Nov 22. PMID 37992261
- [Derived] Kluin-Nelemans HC, Hoster E, Hermine O, Walewski J, Geisler CH, Trneny M, Stilgenbauer S, Kaiser F, Doorduijn JK, Salles G, Szymczyk M, Tilly H, Kanz L, Schmidt C, Feugier P, Thieblemont C, Zijlstra JM, Ribrag V, Klapper W, Pott C, Unterhalt M, Dreyling MH. Treatment of Older Patients With Mantle Cell Lymphoma (MCL): Long-Term Follow-Up of the Randomized European MCL Elderly Trial. J Clin Oncol. 2020 Jan 20;38(3):248-256. doi: 10.1200/JCO.19.01294. Epub 2019 Dec 5. PMID 31804876
- [Derived] Hoster E, Klapper W, Hermine O, Kluin-Nelemans HC, Walewski J, van Hoof A, Trneny M, Geisler CH, Di Raimondo F, Szymczyk M, Stilgenbauer S, Thieblemont C, Hallek M, Forstpointner R, Pott C, Ribrag V, Doorduijn J, Hiddemann W, Dreyling MH, Unterhalt M. Confirmation of the mantle-cell lymphoma International Prognostic Index in randomized trials of the European Mantle-Cell Lymphoma Network. J Clin Oncol. 2014 May 1;32(13):1338-46. doi: 10.1200/JCO.2013.52.2466. Epub 2014 Mar 31. PMID 24687837
- [Derived] Pott C, Hoster E, Delfau-Larue MH, Beldjord K, Bottcher S, Asnafi V, Plonquet A, Siebert R, Callet-Bauchu E, Andersen N, van Dongen JJ, Klapper W, Berger F, Ribrag V, van Hoof AL, Trneny M, Walewski J, Dreger P, Unterhalt M, Hiddemann W, Kneba M, Kluin-Nelemans HC, Hermine O, Macintyre E, Dreyling M. Molecular remission is an independent predictor of clinical outcome in patients with mantle cell lymphoma after combined immunochemotherapy: a European MCL intergroup study. Blood. 2010 Apr 22;115(16):3215-23. doi: 10.1182/blood-2009-06-230250. Epub 2009 Dec 23. PMID 20032498
- See also: official webpage of the European MCLNetwork — http://www.european-mcl.net